CLINICAL TRIAL: NCT03540875
Title: Comparison Between Manual Versus Closed-loop Titration of Propofol and Remifentanil Guided by the qCon and qNox Indexes During Induction and Maintenance of General Anesthesia in Adult Patients: a Multicentre Randomized Controlled Study
Brief Title: Automated Anesthesia Guided by the Conox Monitor for Surgery
Acronym: Conox-loop
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Modification of the device
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/04
Record Dates: First submitted 2018-05-06; First posted 2018-05-30 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Anesthesia, General
Keywords: Anesthesia, general; Total intravenous anesthesia; Closed loop anesthesia; Conox; EEG monitoring; qCon; qNox
MeSH Terms: interventions — Propofol; Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full automation group (Experimental): Full automation control of propofol and remifentanil
  Interventions: Device: Closed loop anesthesia; Drug: Propofol; Drug: Remifentanil
- Control group (Other): Manual control of of propofol and remifentanil using TCI system
  Interventions: Drug: Propofol; Drug: Remifentanil

INTERVENTIONS:
Device: Closed loop anesthesia — Propofol and Remifentanil are administered automatically using a closed-loop system.
  The goal of this study is to compare manual titration versus automated titration of propofol and remifentanil in adult patients undergoing surgery guided by the electro-cortical activity. The aim in both group is to maintain the qCon in the range 40-60 during induction and maintenance of general anesthesia using the propofol in TCI mode. But also the qNox in the range 40-60 using remifentanil. The controller is based on a Proportional-Integral-derivative algorithm which steers a target to the pumps during induction and maintenance of general anesthesia.
  Arms: Full automation group
Drug: Propofol — The dosage is modified automatically by the device or according to the new medical prescription.
Drug: Remifentanil — The dosage is modified automatically by the device or according to the new medical prescription.

SUMMARY:
This study compares automated administration of propofol and remifentanil versus manual administration during general anesthesia for a surgery. The closed-loop coadministration of propofol and remifentanil is guided by qCon and qNox indexes from the Conox monitor.

DETAILED DESCRIPTION:
Several monitors are currently proposed to evaluate the depth of hypnosis. The Conox monitor differentiates itself from the other brain monitor by calculating two EEG indexes, the qCon and the qNox. The qCon corresponds to the depth of the sedation and the qNox relates to the probability that a nociceptive stimulation triggers a movement of the patient. A controller allowing the automated titration of propofol guided by the qCon and remifentanil guided by the qNox has been developed. In preparation for a large multi-center control trial, this prospective randomized study evaluates the effectiveness of such a closed-loop anesthesia system. Two groups of patients are compared: one arm in which propofol and remifentanil are administered by the anesthesiologist using target-controlled infusion (TCI) systems, and the second arm in which propofol and remifentanil are administered automatically by the combined closed-loop anesthesia system. In both groups, the goal is to maintain qCon between 40 and 60, the recommended range during anesthesia by the manufacturer. It is expected the combined closed-loop anesthesia system group to do similar or better control to maintain the qCon in the desired range.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled surgery for at least one hour
* Consent for participation
* Affiliation to the social security system

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients for which Conox monitor should not be used
* Allergies to propofol or remifentanil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Adequate sedation | Start of general anesthesia maintenance, i.e. qCon below 60 for 30 consecutive seconds for the first time, until the end of propofol et remifentanil infusion
  Percentage of time with qCon index within the 40-60 range as recommended by the manufacturer of Conox monitor.
  Data from the Conox monitor (signal quality index, qCon index, qNox index, Suppression ratio) are recorded every second.

SECONDARY OUTCOMES:
Adequate analgesia | Start of general anesthesia maintenance, i.e. qNox below 60 for 30 consecutive seconds for the first time, until the end of propofol et remifentanil infusion
  Percentage of time with qNox index within the 40-60 range as recommended by the manufacturer of Conox monitor.
Occurrence of Burst Suppression Ratio (bsr) | Intraoperative period
  Presence of Burst Suppression defined by a rate > 10% for at least one minute
Dose of hypnotic drug | Intraoperative period
  Total amount of propofol during the induction and the maintenance of the anesthesia
Dose of analgesic drug | Intraoperative period
  Total amount of remifentanil during the induction and the maintenance of the anesthesia
Medical interventions on the dosage of drugs | Intraoperative period
  Number of modifications of target of propofol and remifentanil
Hemodynamic status | Intraoperative period
  Number of episodes of hemodynamic anomalies having required a treatment
Fluid therapy | Intraoperative period
  Intraoperative volume loading and transfusion
Delay before awakening | 12 hours
  Delay between the cessation of infusion of propofol and remifentanil and extubation
Explicit memorization | 48 hours
  Awareness standardized questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hôpital Foch
Locations (3):
- France (3):
  - Service d'Anesthésie Réanimation Chirurgicale, CHU Besançon, Besançon, Bourgogne-Franche-Comté
  - Service d'Anesthésie du Centre Clinical, Soyaux, Poitou-Charentes
  - Service d'Anesthésie, Hôpital Foch, Suresnes, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu N, Chazot T, Hamada S, Landais A, Boichut N, Dussaussoy C, Trillat B, Beydon L, Samain E, Sessler DI, Fischler M. Closed-loop coadministration of propofol and remifentanil guided by bispectral index: a randomized multicenter study. Anesth Analg. 2011 Mar;112(3):546-57. doi: 10.1213/ANE.0b013e318205680b. Epub 2011 Jan 13. PMID 21233500
- [Result] Jensen EW, Valencia JF, Lopez A, Anglada T, Agusti M, Ramos Y, Serra R, Jospin M, Pineda P, Gambus P. Monitoring hypnotic effect and nociception with two EEG-derived indices, qCON and qNOX, during general anaesthesia. Acta Anaesthesiol Scand. 2014 Sep;58(8):933-41. doi: 10.1111/aas.12359. Epub 2014 Jul 4. PMID 24995461